CLINICAL TRIAL: NCT02304263
Title: Assessing Tenofovir Pharmacology in Older HIV Infected Individuals Receiving Tenofovir-based Antiretroviral Therapy
Brief Title: Tenofovir Pharmacology in Older HIV Infected Individuals
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 14-1297; UL1TR001082 (NIH)
Record Dates: First submitted 2014-11-12; First posted 2014-12-01 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: HIV; Aging
Keywords: tenofovir; aging; renal function; HIV; frailty
MeSH Terms: conditions — Frailty | interventions — Iohexol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Younger (18-35 years old): iohexol
  Interventions: Drug: iohexol
- Older (>60 years old): iohexol
  Interventions: Drug: iohexol

INTERVENTIONS:
Drug: iohexol — 5mL bolus of 300 mg/ml iohexol (Omnipaque) over 2 minutes
  Other Names: Omnipaque

SUMMARY:
Tenofovir continues to play a vital role in the treatment of the human immunodeficiency virus (HIV) and as the age of the HIV-infected population increases in the United States and worldwide, there is an urgent need to understand the extent to which older age influences the way this antiretroviral medication works in the body. The investigators study aims to characterize and compare the pharmacology of tenofovir in older versus younger HIV-infected adults and to assess kidney function over the course of approximately one year. The investigators will be analyzing tenofovir levels in different compartments of the blood and in hair samples, and will be assessing the relationship between tenofovir concentrations and changes in kidney function over time in the older and younger cohorts. Lastly, the investigators will be evaluating the relationship between tenofovir concentrations and functional status (including body composition, bone mineral density, and frailty) in study participants.

DETAILED DESCRIPTION:
Despite a growing population of older HIV infected persons world-wide, major knowledge gaps exist with regards to the pharmacokinetics and pharmacodynamics of antiretroviral drugs in older persons. In the United States, the median age of HIV-infected persons is expected to surpass 50 years by 2015. A global report from UNAIDS indicated that for the first time since the start of the HIV epidemic, 10% of the adult population currently living with HIV in low- and middle-income countries is aged 50 or older, and in high-income countries, approximately 30% of adults living with HIV are aged 50 years and over. Hypertension, diabetes, cardiovascular disease, cancer, osteoporosis, cognitive decline, and hepatic and renal dysfunction are commonly encountered problems in older persons. Frailty is also commonly encountered in the aging population and is defined as the cumulative effects of age-related declines in multiple physiological systems and homeostatic mechanisms, resulting in greater vulnerability to stressors. People living with HIV have a higher prevalence and earlier onset of age-related declines in health, including frailty, compared to HIV-uninfected adults. The emphasis of HIV management over the past decade has shifted from the prevention of AIDS complications, to the management of chronic non-infectious comorbidities in an increasingly older and more complicated patient population. Age-related declines in health along with established changes in body composition as individuals get older (increased body fat, decreased lean mass), may impact the pharmacokinetics of antiretroviral medications used in the treatment of HIV, but this has not been studied adequately. To date, there is a substantial lack of information regarding the pharmacokinetics of antiretroviral medications, including tenofovir (TFV), in older HIV-infected adults. As evidence, the 'Geriatric Use' sections of the Viread® (tenofovir disoproxil fumarate, TDF)-containing products state the following, "Clinical studies of Viread® did not include sufficient numbers of subjects aged 65 and over to determine whether they respond differently from younger subjects. In general, dose selection for the elderly patient should be cautious, keeping in mind the greater frequency of decreased hepatic, renal, or cardiac function, and of concomitant disease or other drug therapy." These gaps in knowledge arise from underrepresentation of older individuals in the early phases of drug development. This is especially true for antiretroviral drugs because HIV-infection afflicted mostly young people at the time most antiretroviral drugs were being developed. It is important to realize that HIV-infected individuals are now reaching older ages in high numbers, and that studies are urgently needed to optimize drug responses in this population. A major gap in knowledge is the lack of information surrounding the association between functional (frailty) status and the pharmacology of antiretroviral medications in older HIV-infected individuals.

As older adults experience natural declines in renal function, drugs that are renally eliminated may accumulate in the systemic circulation, thus increasing the risk for toxicities. Tenofovir is renally eliminated and its principal dose-related toxicity is new or worsening renal impairment, meaning that slowed elimination may accelerate damage to the kidneys in this population. In order to assess changes in renal function clinically, regression equations that incorporate age, such as Cockgroft-Gault and MDRD, are utilized, but depend on serum creatinine (endogenous muscle byproduct). Serum creatinine is not an ideal marker in older populations because muscle mass decreases with age. A better method to quantify actual GFR is by evaluating the plasma clearance of the contrast agent, iohexol (iGFR). This approach is considered a gold standard for assessing renal function at all ages.

The Anderson Laboratory recently validated a method for measuring the intracellular concentration of tenofovir-di-phosphate (TFV-DP), the active form of tenofovir, in red blood cells (RBC) using dried blood spots (DBS )to indicate both recent and cumulative dosing. Similar to the benefits provided by hemoglobin A1C testing in diabetes therapy, TFV-DP in DBS testing allows for a much needed quantitative approach for assessing cumulative exposure to tenofovir over long periods of time. This is enabled by the 17 day half-life for TFV-DP in RBC. Measuring TFV concentrations in scalp hair is an alternative method for measuring cumulative exposure to the drug over long periods of time (weeks to months), as demonstrated by researchers at the University of California San Francisco.

These novel biomarkers for long-term tenofovir exposure provide an opportunity to compare cumulative tenofovir exposure in older versus younger individuals. Long-term use of tenofovir is associated with two main adverse effects, namely changes in bone mineral density and renal function, however the link between age, tenofovir exposure, and rate of decline in bone mineral density and renal function have not been fully elucidated. The goals of the present study are to characterize and compare the pharmacokinetics of TFV in older HIV-infected adults versus younger HIV-infected adults and to assess the changes in bone mineral density and renal function (using iohexol) over an approximate one year time period in these two cohorts. The study will also include measures of body composition (using duel-energy x-ray absorptiometry, DXA) and functional status (frailty) and will assess the relationships between these factors and TFV pharmacology in both the younger and older HIV-infected cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be between either 18-30 years or >60 years of age
2. Participants must be HIV-positive and receive care from the Infectious Disease (IDGP) Clinic at the University of Colorado Hospital
3. Participants must have a history of consistent antiretroviral therapy with a qualifying regimen that includes TFV for at least one year
4. Participants must have a suppressed HIV-RNA load (<48 copies/mL on consecutive visits) while on a TFV-based regimen

Exclusion Criteria:

1. eGFR < 50 ml/min/1.73 m2
2. Use of concomitant nephrotoxic agents (aminoglycosides, amphotericin, cyclosporine, etc.)
3. Allergy to iodine and/or iohexol
4. Uncontrolled, un-medicated hyperthyroidism
5. Plans to relocate out of state in the next year
6. Currently pregnant or plans to become pregnant in the next year, currently breastfeeding
7. Weight ≥ 300 lbs
8. Bilateral hip replacements, bilateral hip pins or screws, metallic rods or spinal fusion devices in the lumbar spine
9. Any medical, social, or mental-health issue(s) that, in the opinion of the investigators, could interfere with the study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1 participants will include 22 adults between the ages of 18-35 years and Group 2 will include 22 individuals >60 years old.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
iGFR values and pharmacokinetic parameters of TFV in plasma, RBC, DBS, peripheral blood mononuclear cells (PBMC), and scalp hair in older versus younger adults | 1 year
iGFR change over a one year time period in older versus younger adults | 1 year
Bone mineral density DXA score changes for hip and lumbar vertebrae over a one year time period in older versus younger adults | 1 year
Relationship between TFV pharmacology, iGFR,and frailty score in older versus younger adults | 1 year

SECONDARY OUTCOMES:
Clinical and laboratory predictors of iGFR and TFV levels in blood and hair, including genetic predictors in those who consent, in older versus younger adults | 1 year
Pharmacological measures of cumulative drug exposure in relation to traditional measures of drug adherence in older versus younger adults (Compare DBS and hair drug levels to pharmacy refill data and self-report (using visual analog scale).) | 1 year
  Compare DBS and hair drug levels to pharmacy refill data and self-report (using visual analog scale).
Estimated GFR (using Cockgroft-Gault, MDRD, and CKD-Epi) values versus iGFR values in older versus younger adults | 1 year
Amount of muscle and fat mass (determined by DXA body composition scan) in older versus younger adults | 1 year
Pharmacokinetic parameters, including steady-state concentrations, of antiretroviral drugs other than tenofovir in older versus younger adults | 1 year
  Measurement of the volumes of distribution (Vd) and elimination rate constants (ke) will be used in the determination of steady-state concentrations.
Panel of immune activation and inflammation markers in older versus younger adults | 1 year
  Panel includes: HLA-DR, CD38, CD28, CD14, CD27, IL-6, TNF-1 and -2 receptors
Endogenous nucleotide pools in older versus younger adults | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sharon M Seifert, PharmD, Principal Investigator — University of Colorado, Denver